CLINICAL TRIAL: NCT02372292
Title: Value of Renal Vascular Doppler Sonography in Management of Decompensated Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Özgür Ulaş Özcan, MD, Ankara University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Ankararenal
Record Dates: First submitted 2015-02-13; First posted 2015-02-26 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Cardiorenal Syndrome
Keywords: cardiorenal syndrome, decompensated heart failure, renal resistivity index, venous impedance index, kidney failure
MeSH Terms: conditions — Cardio-Renal Syndrome; Renal Insufficiency | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Patients with type 1 cardiorenal syndrome who had improvement of renal functions along with diuretic therapy. Intravenous furosemide treatment.
  Interventions: Drug: intravenous furosemide
- Group 2 (Active Comparator): Patients with type 1 cardiorenal syndrome who did not have improvement of renal functions along with diuretic therapy. Intravenous furosemide treatment.
  Interventions: Drug: intravenous furosemide

INTERVENTIONS:
Drug: intravenous furosemide — Decongestant therapy for decompensated heart failure which may be administrated as intravenous bolus or infusion
  Other Names: Lasix

SUMMARY:
Although the traditional determinant of renal dysfunction in heart failure was suggested as decreased cardiac output and renal hypo perfusion, recent studies have demonstrated the association of persistent systemic venous congestion and kidney dysfunction. Relief of the congestion has demonstrated to improve renal functions in decompensated heart failure. The current trial was set up to investigate the changes of renal venous impedance and renal arteriolar resistivity indices with diuretic therapy, in patients with congestive renal failure. The investigators asked whether measurement of renal venous impedance index or renal arteriolar resistivity index can guide the practice of diuretic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated heart failure
* Elevated serum creatinine levels on admission

Exclusion Criteria:

* Atrial fibrillation
* Obstructive uropathy
* Patients with ascites
* Patients who exposed the potential nephrotoxic drugs in the previous week (metformin, antibiotics, chemotherapeutics, iodinated contrast agents and non-steroidal anti-inflammatory agents)
* Patients who needed positive inotropic agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Alterations in the renal arterial resistivity index | during hospitalization, an expected average of 4 weeks.
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.

SECONDARY OUTCOMES:
Alterations in the renal venous impedance index | during hospitalization, an expected average of 4 weeks.
  Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School Of Medicine, Department of Cardiology, Ankara, Turkey (Türkiye)